CLINICAL TRIAL: NCT02976935
Title: FUNCTIONAL MAGNETIC RESONANCE LUNG IMAGING USING INHALED HYPERPOLARISED 129Xe
Brief Title: Functional MR Lung Imaging Using Hyperpolarised 129Xe
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 13104
Record Dates: First submitted 2016-02-09; First posted 2016-11-30 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: COPD; IPF
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Subjects will receive 1L non-hyperpolarised 129Xenon to inhale. Then:Subjects will inhale the first hyperpolarised 129Xenon calibration dose (up to 1L, which may be a mix of hyperpolarised 129Xenon and N2) and hold their breath while the MRI scan is performed. Then:A further series of inhalations will be performed up to a maximum of 3 (maximum total exposure to hyperpolarised 129Xenon will be 3.6L). Optional Study Visit #2:Identical to Study Visit 1 but with the further series of inhalations being up to a maximum of 4 (maximum total exposure to hyperpolarised 129Xenon will be 5L).Optional Study Visit #3: Identical to Study Visit 2 (maximum total exposure to hyperpolarised 129Xenon will be 5L)
  Interventions: Other: hyperpolarised 129 Xenon
- Chronic Obstructive Pulmonary Disease: Subjects will receive 1L bag of non-hyperpolarised 129Xenon to inhale. Then:Subjects will inhale the first hyperpolarised 129Xenon calibration dose (up to 1L, which may be a mix of hyperpolarised 129Xenon and N2) and hold their breath for required time while the MRI scan is performed.Then:A further series of inhalations will be performed up to a maximum of 3 (maximum total exposure to hyperpolarised 129Xenon will be 3.6L). Optional Study Visit #2: Identical to Study Visit 1 (maximum total exposure to hyperpolarised 129Xenon will be 3.6L)
  Interventions: Other: hyperpolarised 129 Xenon

INTERVENTIONS:
Other: hyperpolarised 129 Xenon — Hyperpolarised 129 Xe to assess lung function

SUMMARY:
The aim of this study is to investigate the potential value of a novel imaging technique (hyperpolarized 129Xe lung imaging) in the diagnosis and assessment of lung disease in patients with COPD and IPF.

ELIGIBILITY:
General Inclusion criteria

* Male or Female aged over 18 years.
* Capacity to give informed consent
* Normal blood pressure (systolic BP > 100 mmHg and diastolic BP > 70 mmHg)
* Resting heart rate > 50 bpm
* For women, negative urinary β-hCG at the screening and subsequent visits
* Subject able to hold breath for 10 seconds
* Subject able to fit into 129Xe chest coil used for MRI
* Subject able to understand the requirements of the study and to cooperate with the study procedures

Inclusion criteria

HEALTHY VOLUNTEERS

• No significant respiratory disease within the last year

PATIENTS

COPD

* Evidence of airflow obstruction (FEV/FVC <0.7) and FEV1 <80% predicted post bronchodilator
* Minimum FVC 1.5L

Exclusion criteria

HEALTHY VOLUNTEERS

* Unsuitable for MRI scanning (e.g. have metal implants or pacemaker or contraindicated following questionnaire)
* Acute respiratory illness within 30 days of MRI
* Subject has received an IMP (not including hyperpolarized 129Xe) within 30 days of MRI and administration of 129Xe deemed inappropriate in context of other study
* Subject deemed unlikely to comply with instructions during imaging
* Do not meet the inclusion criteria above
* Subject not deemed fit enough to tolerate procedure
* Subject deemed unsuitable by clinical investigator for other reasons

PATIENTS

* Unsuitable for MRI scanning (e.g. have metal implants or pacemaker or contraindicated following questionnaire)
* Acute respiratory illness within 30 days of MRI
* Subject has received an IMP (not including hyperpolarized 129Xe) within 30 days of MRI and administration of 129Xe deemed inappropriate in context of other study
* Subject deemed unlikely to comply with instructions during imaging
* Do not meet the inclusion criteria above
* Subject not deemed fit enough to tolerate procedure
* Subject deemed unsuitable by clinical investigator for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers, COPD
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-02; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Acquisition of baseline data and images to investigate use of hp129Xe as a diagnostic tool | 4 years
  i) Obtain baseline data for each group with matched clinical data (e.g. pulmonary function tests) allowing comparison with existing clinical diagnostic techniques and also determining correlation with disease severity ii) Use the images obtained to set up standard sequencing protocols and define algorithms and inform power calculations for subsequent studies

SECONDARY OUTCOMES:
Collation of data regarding ability of participants to adhere to the study protocol | 4 years
  1) To collate data regarding the ability of participants of each group to adhere to the protocol thus informing the study design of future trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Hyperpolarised Imaging Lung Facility, QMC, Uni of Nottingham, Nottingham, United Kingdom